CLINICAL TRIAL: NCT02339363
Title: Differential Effects of Sitting Meditation and Hatha Yoga on Working Memory, Stress, and Mindfulness Among Adolescents in a School Setting
Brief Title: Effects of Sitting Meditation and Hatha Yoga in Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliant International University (Other)
Responsible Party: Principal Investigator, Kristen Jastrowski Mano, Assistant Professor, Alliant International University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Quach-1-2013
Record Dates: First submitted 2015-01-09; First posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Anxiety; Psychological Stress
Keywords: mindfulness; adolescents; working memory; stress; anxiety
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sitting Meditation (Experimental): 4 weeks (45-min sessions, 2x per week) of sitting meditation, based on MBSR. The sitting meditation condition consisted of three parts: (a) breathing techniques, (b) meditation, and (c) discussion. Participants in the sitting meditation group learned new types of sitting meditation each week. Participants in the sitting meditation group received a CD that consisted of audio meditations that they could follow along at home. The sitting meditation participants were encouraged to practice formal sitting meditation for 15 to 30 minutes every day and asked to record details of their practice on their daily home practice logs.
  Interventions: Behavioral: Sitting Meditation
- Hatha Yoga (Experimental): 4 weeks(45-min sessions, 2x per week) of Hatha Yoga. The adolescent hatha yoga curriculum was used with permission from Shanti Generation Yoga © (2009) created by Abby Wills. The hatha yoga sessions consisted of three parts: (a) breathing techniques, (b) yoga poses, and (c) discussion. Participants in the hatha yoga group learned a series of new yoga poses each week, as well as reviewed old poses. During the first session, participants in the hatha yoga group received a DVD that contained five yoga lessons corresponding to the yoga poses being taught in the intervention. Participants were encouraged to practice the series of yoga poses at home for 15 to 30 minutes each day and record their home practice in their daily home practice logs.
  Interventions: Behavioral: Hatha yoga
- Waitlist Control (No Intervention): 4-week waitlist control condition. Completed all study measures at same time points as experimental groups. Were randomly assigned to one of the two active treatment conditions after completing the waitlist period.

INTERVENTIONS:
Behavioral: Sitting Meditation — 4 weeks Sitting Meditation
  Arms: Sitting Meditation
Behavioral: Hatha yoga — 4 weeks of Hatha yoga
  Arms: Hatha Yoga

SUMMARY:
The present study was a randomized controlled trial that explored the feasibility, acceptability, and effectiveness of short-term mindfulness training among adolescents. The primary purpose was to investigate the effectiveness of two main Mindfulness-Based Stress Reduction components-sitting meditation and hatha yoga-on working memory, stress, anxiety and mindfulness. The influence of daily home practice compliance on intervention outcomes was also examined.

DETAILED DESCRIPTION:
The present study was a randomized controlled trial that explored the feasibility, acceptability, and effectiveness of short-term mindfulness training among adolescents. The primary purpose was to investigate the effectiveness of two main Mindfulness-Based Stress Reduction components-sitting meditation and hatha yoga-on working memory, stress, anxiety and mindfulness. The influence of daily home practice compliance on intervention outcomes was also examined. Participants (N = 198 adolescents) were recruited from a large public middle school in southern California. Participants were randomly assigned to sitting meditation, hatha yoga, or a waitlist control group. Participants were asked to complete a computerized working memory task, and self-report measures of perceived stress, anxiety, and mindfulness at pre- and post-intervention/waitlist, as well as one-month follow-up. A series of mixed-design analyses of variance (ANOVAs) were used to examine changes in working memory, stress, anxiety, and mindfulness between groups at pre- and post- intervention.

ELIGIBILITY:
Inclusion Criteria:

* Students currently enrolled in school
* Between the ages of 12 - 17 years old
* English speaking-to understand and complete the measures
* Able to attend the weekly hatha yoga or sitting meditation sessions
* Not reporting any injuries or health condition(s) that might limit their physical activity

Exclusion Criteria:

* hearing impairments, injuries, or physical disabilities that would hinder them from fully participating in intervention

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 198 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Working Memory Capacity: Automated Operational Span Task (AOSPAN) | pre-intervention and post-intervention (waitlist), t the end of the 4-week intervention (waitlist) period
  Participants completed the AOSPAN prior to beginning their group condition (sitting meditation, Hatha yoga, or waitlist control) and again at the end of the 4-week intervention (waitlist) period.

SECONDARY OUTCOMES:
Stress: Perceived Stress Scale (PSS-10) | pre-intervention and post-intervention (waitlist), t the end of the 4-week intervention (waitlist) period
  Participants completed the PSS-10 prior to beginning their group condition (sitting meditation, Hatha yoga, or waitlist control) and again at the end of the 4-week intervention (waitlist) period.
Anxiety: Screen for Child Anxiety and Related Emotional Disorders (SCARED) | pre-intervention and post-intervention, t the end of the 4-week intervention (waitlist) period
  Participants completed the SCARED prior to beginning their group condition (sitting meditation, Hatha yoga, or waitlist control) and again at the end of the 4-week intervention (waitlist) period.
Mindfulness: Child Acceptance and Mindfulness Measure (CAMM) | pre-intervention and post-intervention (waitlist), t the end of the 4-week intervention (waitlist) period
  Participants completed the CAMM prior to beginning their group condition (sitting meditation, Hatha yoga, or waitlist control) and again at the end of the 4-week intervention (waitlist) period.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Jastrowski Mano, Ph.D., Principal Investigator — Alliant International University

REFERENCES:
- [Derived] Quach D, Jastrowski Mano KE, Alexander K. A Randomized Controlled Trial Examining the Effect of Mindfulness Meditation on Working Memory Capacity in Adolescents. J Adolesc Health. 2016 May;58(5):489-96. doi: 10.1016/j.jadohealth.2015.09.024. Epub 2015 Nov 11. PMID 26576819